CLINICAL TRIAL: NCT01279928
Title: Detection of Vascular Injury in Diabetes Through Eye and Nailfold Data (DIVIDEND) - A Pilot Study
Acronym: DIVIDEND
Status: Completed | Type: Observational
Sponsor: John Hunter Hospital (Other Government)
Responsible Party: Associate Professor Glenn Reeves, John Hunter Hospital
Other Study IDs: HNEHREC 09/04/15/5.10
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: paediatric and adolescent population; nailfold capillaroscopy; laser Doppler flowmetry; retinal vessel calibre; retinal vessel fractal analysis; 24 hour Ambulatory Blood Pressure Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Pressure Monitors; Laser-Doppler Flowmetry

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 1 Diabetes Paediatric: Paediatric patients aged 8-18 with diagnosed Diabetes Mellitis Type 1 attending paediatric clinic at John Hunter Hospital.
  Interventions: Procedure: Video Nailfold Capillaroscopy; Device: Ambulatory 24 hr Blood Pressure Monitoring; Procedure: Fundoscopy of eyes; Procedure: Laser Doppler Flowmetry

INTERVENTIONS:
Procedure: Video Nailfold Capillaroscopy — Single session of video Nailfold Capillaroscopy wit KKK technology
Device: Ambulatory 24 hr Blood Pressure Monitoring — 24 hr upper arm cuff measurement of Blood Pressure
Procedure: Fundoscopy of eyes — examination of microvascular health of eye with the use of opthalmoscope
Procedure: Laser Doppler Flowmetry — Examination of vascular flow

SUMMARY:
This project aimed to explore novel methods of detecting small blood vessel disease in a paediatric population with type 1 diabetes mellitus. To do this the techniques of Nailfold capillaroscopy, laser Doppler flowmetry, retinal (eye) vessel analysis and 24-hr Ambulatory Blood Pressure Monitoring were used. Each of these techniques investigated different areas of small blood vessels around the body.

It was hypothesized that in a paediatric population with type 1 diabetes mellitus the novel investigations would be associated with small blood vessel disease and that widespread changes to these blood vessels would be detected through associations between the different novel investigations.

ELIGIBILITY:
Inclusion Criteria:

* 8-18 years old
* Have a diagnosis of type 1 diabetes mellitus

Exclusion Criteria:

* < 8 years or > 18 years old
* Significant autoimmune rheumatological disease (e.g. lupus or dermatomyositis)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants were recruited from the John Hunter Children's Hospital paediatric diabetes clinic. They were between the ages of 8-18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rani Bhatia, MD, Principal Investigator — John Hunter Children's Hospital
Locations (1):
- John Hunter Children's Hospital, New Lambton, New South Wales, Australia

REFERENCES:
- [Derived] Hosking SP, Bhatia R, Crock PA, Wright I, Squance ML, Reeves G. Non-invasive detection of microvascular changes in a paediatric and adolescent population with type 1 diabetes: a pilot cross-sectional study. BMC Endocr Disord. 2013 Oct 5;13:41. doi: 10.1186/1472-6823-13-41. PMID 24093770